CLINICAL TRIAL: NCT04141228
Title: Evaluation of Hospital Healthcare Utilization and Costs Among Hospitalized Venous Thromboembolism (VTE) Patients Treated With Apixaban or Warfarin in the United States
Brief Title: A Study of Hospital Healthcare Use and Cost in Patients in the Hospital With a Venous Thromboembolism (VTE) Treated With Apixaban or Warfarin in the US
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-589
Record Dates: First submitted 2019-10-21; First posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Venous Thromboembolism (VTE)
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients receiving apixaban: With or without low molecular weight heparin in the inpatient/emergency department (ED) setting
- Patients receiving warfarin: With or without low molecular weight heparin in the inpatient/emergency department (ED) setting

SUMMARY:
A study involving real-world database analysis to evaluate the hospital healthcare utilization and costs, and all-cause, major bleeding-, clinically relevant bleeding-, any bleeding-, and venous thromboembolism (VTE)-related hospital readmissions among hospitalized VTE patients treated with apixaban or warfarin, with or without low molecular weight heparin (LMWH)

ELIGIBILITY:
Inclusion Criteria:

* Have a primary diagnosis of VTE identified by ICD-9-CM or ICD-10 codes from the Premier Hospital database between 01-Aug-2014 and 31-May-2016
* Age 18 years or older as of index hospitalization with VTE diagnosis
* Patients will be required to have received apixaban or warfarin with or without LMWH (index drugs) during the index hospitalizations

Exclusion Criteria:

* Received both apixaban and warfarin during the index hospitalization. This exclusion criterion will allow to cleanly group patients into the apixaban and warfarin usage cohorts.
* Received any other Direct oral anticoagulants (DOAC) including rivaroxaban, dabigatran, and edoxaban during the index hospitalization
* Have any primary or secondary diagnosis code for Atrial fibrillation/Atrial flutter (AF/AFL), or pregnancy, or records of inferior vena cava filter (IVCF) usage during the index hospitalizations or the baseline periods.
* Patients transferred from other facilities

Other protocol-defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients with a hospital or ED discharge International Classification of Diseases, Ninth Revision, Clinical Modification (ICD-9-CM) or ICD-10 code indicating a primary diagnosis of VTE identified from the Premier Hospital database between 01-Aug-2014 and 31-May-2016. Patients who received apixaban or warfarin with or without LMWH during any time of the hospitalization (from admission to discharge) will be identified. Patients receiving both apixaban and warfarin, or any other direct oral anticoagulant (DOAC), including rivaroxaban, dabigatran, and edoxaban, during the index hospitalizations will be excluded from the study population. Patients will be required to have no evidence of atrial fibrillation (AF) or atrial flutter (AFL) during the index hospitalizations or the baseline periods.
Sampling Method: Probability Sample
Enrollment: 28000 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Hospital Length of stay (LOS) | During the index hospitalization (Up to 30 days)
Hospital cost | During the index hospitalization (Up to 30 days)

SECONDARY OUTCOMES:
Proportion of patients with major bleeding (MB)-related hospital readmissions | During 1 month after the index hospitalization
Proportion of patients with clinically relevant bleeding (CRB)-related hospital readmissions | During 1 month after the index hospitalization
Proportion of patients with any bleeding-related hospital readmissions | During 1 month after the index hospitalization
Proportion of patients with VTE-related hospital readmissions | During 1 month after the index hospitalization
Proportion of patients with combined VTE- or MB-related hospital readmissions | During 1 month after the index hospitalization
Proportion of patients with all-cause hospital readmissions | During 1 month after the index hospitalization
Hospital Length of stay (LOS) for major bleeding-related hospital readmissions | During 1 month following the VTE hospitalization
Hospital costs of readmissions for major bleeding-related hospital readmissions | During 1 month following the VTE hospitalization
Hospital charges of readmissions for major bleeding-related hospital readmissions | During 1 month following the VTE hospitalization]
Mean number of hospital readmissions for major bleeding-related hospital readmissions | During 1 month following the VTE hospitalization
Hospital LOS for clinically relevant bleeding-related hospital readmissions | During 1 month following the VTE hospitalization
Hospital costs of readmissions for clinically relevant bleeding-related hospital readmissions | During 1 month following the VTE hospitalization
Hospital charges of readmissions for clinically relevant bleeding-related hospital readmissions | During 1 month following the VTE hospitalization
Mean number of hospital readmissions for clinically relevant bleeding-related hospital readmissions | During 1 month following the VTE hospitalization
Hospital LOS for any bleeding-related hospital readmissions | During 1 month following the VTE hospitalization
Hospital costs of readmissions for any bleeding-related hospital readmissions | During 1 month following the VTE hospitalization
Hospital charges of readmissions for any bleeding-related hospital readmissions | During 1 month following the VTE hospitalization
Mean number of hospital readmissions for any bleeding-related hospital readmissions | During 1 month following the VTE hospitalization
Hospital LOS for VTE-related hospital readmissions | During 1 month following the VTE hospitalization
Hospital costs of readmissions for VTE-related hospital readmissions | During 1 month following the VTE hospitalization
Hospital charges of readmissions for VTE-related hospital readmissions | During 1 month following the VTE hospitalization
Mean number of hospital readmissions for VTE-related hospital readmissions | During 1 month following the VTE hospitalization
Hospital LOS for combined VTE- or MB-related hospital readmissions | During 1 month following the VTE hospitalization
Hospital costs of readmissions for combined VTE- or MB-related hospital readmissions | During 1 month following the VTE hospitalization
Hospital charges of readmissions for combined VTE- or MB-related hospital readmissions | During 1 month following the VTE hospitalization
Mean number of hospital readmissions for combined VTE- or MB-related hospital readmissions | During 1 month following the VTE hospitalization
Hospital LOS for all-cause hospital readmissions | During 1 month following the VTE hospitalization
Hospital costs of readmissions for all-cause hospital readmissions | During 1 month following the VTE hospitalization
Hospital charges of readmissions for all-cause hospital readmissions | During 1 month following the VTE hospitalization
Mean number of hospital readmissions for all-cause hospital readmissions | During 1 month following the VTE hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Flemington, New Jersey, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm